CLINICAL TRIAL: NCT02289027
Title: A Phase I/II Double-blind, Randomized, Placebo Controlled, Safety and Immunogenicity, Dose-finding Trial of the Monovalent Zaire Ebola Chimpanzee Adenovirus Vector Candidate Vaccine cAd3-EBOZ in Healthy Adults in Switzerland
Brief Title: A Clinical Trial on the Candidate Vaccine cAd3-EBOZ in Healthy Adults in Switzerland
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Infectious Disease Service, CHUV, Lausanne (Unknown); Center for Primary Care and Public Health (Unisante), University of Lausanne, Switzerland (Other); University of Lausanne Hospitals (Other); Swiss Tropical & Public Health Institute (Other); University of Lausanne (Other); GlaxoSmithKline (Industry); World Health Organization (Other); Immunology and Allergy Service, CHUV, Lausanne (Unknown)
Responsible Party: Principal Investigator, François Spertini, Head physician Immunology and Allergy, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: cAd3-EBOZ Lau
Record Dates: First submitted 2014-10-14; First posted 2014-11-13 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Ebola Vaccines
Keywords: Ebola, Ebolavirus
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Deployed volunteers - Group 1 (Experimental): Low dose cAd3-EBOZ (2.5x10e10 vp)
  Interventions: Biological: cAd3-EBOZ vaccine
- Deployed volunteers - Group 2 (Experimental): High dose cAd3-EBOZ (5x10e10 vp)
  Interventions: Biological: cAd3-EBOZ vaccine
- Not deployed volunteers - Group 3 (Experimental): Low dose cAd3-EBOZ (2.5x10e10 vp)
  Interventions: Biological: cAd3-EBOZ vaccine
- Not deployed volunteers - Group 4 (Experimental): High dose cAd3-EBOZ (5x10e10 vp)
  Interventions: Biological: cAd3-EBOZ vaccine
- Not deployed volunteers - Group 5 (Placebo Comparator)
  Interventions: Biological: Placebo (for cAd3-EBOZ vaccine)

INTERVENTIONS:
Biological: cAd3-EBOZ vaccine
  Arms: Deployed volunteers - Group 1; Deployed volunteers - Group 2; Not deployed volunteers - Group 3; Not deployed volunteers - Group 4
Biological: Placebo (for cAd3-EBOZ vaccine) — Diluent
  Arms: Not deployed volunteers - Group 5

SUMMARY:
The objective of this trial is to assess in healthy adults the safety and reactogenicity of a new candidate vaccine, cAd3-EBOZ, made of a chimpanzee Adenovirus vector encoding the glycoprotein of Zaire Ebola virus. The secondary objectives will be to assess the immunogenicity of the candidate vaccine and find the most suitable dose for further deployment in epidemic areas in Africa. The 120 planned study subjects will be composed of possibly exposed volunteers owning to organisations such as "Médecins sans frontières" and susceptible to be deployed in the outbreak zone (named as "possibly exposed volunteers"). The other volunteers will be adults with no planned travels to the epidemic zone (named as "not exposed volunteers"). The first group will be randomly allocated to two different groups (low dose = single injection of 2.5x10e10 viral particles (vp), high dose = single injection of 5x10e10 vp). The second group will be randomly allocated to three different groups (low dose = single injection of 2.5x10e10 viral particles (vp), high dose = single injection of 5x10e10 vp or placebo = single injection of vaccine diluent). The design will be double-blind. Follow-up visits will take place at Day 1, 7, 14, 28, 90 and 180.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 18 to 65 years
2. Able and willing (in the Investigator's opinion) to comply with all study requirements
3. Willing to allow the investigators to discuss the volunteer's medical history with their general practitioner
4. For females of reproductive capacity and males, having practiced continuous effective contraception for 21 days prior to enrolment, and willing to practice continuous effective contraception for 3 months post vaccination
5. For females of reproductive capacity, having a negative pregnancy test on the day(s) of screening and vaccination if >7 days interval
6. Agreement to refrain from blood donation during the course of the study
7. Provide written informed consent

Exclusion Criteria:

1. Participation in another research study involving receipt of an investigational product in the 30 days preceding enrolment, or planned use during the study period
2. Prior receipt of an investigational Ebola or Marburg vaccine or a chimpanzee adenovirus vectored vaccine
3. Receipt of any live, attenuated vaccine within 28 days prior to enrolment
4. Receipt of any subunit or killed vaccine within 14 days prior to enrolment (influenza vaccination is encouraged prior to participation)
5. Receipt of any investigational vaccine within 3 months prior to enrollment
6. Administration of immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate
7. Any confirmed or suspected immunosuppressed or immunodeficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressive medication within the past 6 months (inhaled and topical steroids are allowed)
8. History of allergic reactions likely to be exacerbated by any component of the vaccine,
9. Any history of hereditary angioedema, acquired angioedema, or idiopathic angioedema.
10. Any history of anaphylaxis in reaction to vaccination
11. Pregnancy, lactation or willingness/intention to become pregnant during the study
12. History of cancer (except basal cell carcinoma of the skin and cervical carcinoma in situ)
13. History of serious psychiatric condition
14. Poorly controlled asthma or thyroid disease
15. Seizure in the past 3 years or treatment for seizure disorder in the past 3 years
16. Bleeding disorder (eg. Factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following intramuscular injections or venepuncture
17. Any other serious chronic illness requiring hospital specialist supervision
18. Current anti-tuberculosis prophylaxis or therapy
19. Suspected or known current alcohol abuse
20. Suspected or known injecting drug abuse in the 5 years preceding enrolment
21. Seropositive for hepatitis B surface antigen (HBsAg)
22. Seropositive for hepatitis C virus (antibodies to HCV)
23. Any clinically significant abnormal finding on screening biochemistry or haematology blood tests or urinalysis
24. Any other significant disease, disorder or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-10; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Solicited local and systemic reactogenicity signs and symptoms | Daily for 7 days following the vaccination
  Solicited local signs and symptoms include: pain at injection site; erythema at injection site; swelling at injection site. They will be assessed according to a preestablished scale (grade 1 to 3).
  Solicited systemic signs and symptoms include: fever; tachycardia; bradycardia; systolic hypertension; distolic hypertension; systolic hypotension. They will be assessed according to a preestablished scale (grade 1 to 3).
Unsolicited adverse events of all severities | Through 28 days after the vaccination
  Unsolicited adverse events will be assessed according to a severity grading scale (grade 1 to 3).
Change from baseline for safety laboratory measures | Through 6 months after the vaccination
  Safety laboratory measures include: hemoglobin; white blood cells count; neutrophil count; lymphocyte count; platelets; total bilirubin; alanine aminotransferase (ALT); aspartate aminotransferase (AST); alkaline phosphatase; creatinine; urea; sodium; potassium; partial thromboplastin time (aPTT). They will be assessed according to a severity grading scale (grade 1 to 3).
Occurrence of serious adverse events and suspected unexpected serious adverse reactions | Through 6 months after the vaccination
  SAE are defined as AE that result in any of the following outcomes, whether or not considered related to the study intervention:
  * Death
  * Life-threatening event
  * Persistent or significant disability or incapacity
  * Hospitalisation
  * An important medical event (that may not cause death, be life threatening, or require hospitalisation) that may, based upon appropriate medical judgment, jeopardise the volunteer and/or require medical or surgical intervention to prevent one of the outcomes listed above.
  * Congenital anomaly or birth defect.
  A SUSAR is a suspected unexpected serious adverse reaction thought to be possibly, probably or definitely related to an IMP. No category of SAE has been defined as 'expected'.

SECONDARY OUTCOMES:
Antibody responses as measured by ELISA (anti-EBOZ immunoglobulins titers) and by antigen-specific neutralization assays | Through 6 months after the vaccination
T cell immune responses as measured by ex-vivo ELISPOT | Through 6 months after the vaccination

OTHER OUTCOMES:
T cell immune responses as measured by intracellular cytokine staining assays (ICS) | Through 6 months after the vaccination
T cell immune responses as measured by 6-day culture cytokine production by Multiplex and flow cytometry | Through 6 months after the vaccination
HLA typing | On Day 0 (day of vaccination)
Vaccine-induced mRNA expression profiles (transcriptomics) | Through 28 days after the vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Blaise Genton, MD PhD, Principal Investigator — CHUV and PMU
Locations (1):
- Clinical Trial Unit Lausanne, Lausanne, Switzerland

REFERENCES:
- [Derived] De Santis O, Audran R, Pothin E, Warpelin-Decrausaz L, Vallotton L, Wuerzner G, Cochet C, Estoppey D, Steiner-Monard V, Lonchampt S, Thierry AC, Mayor C, Bailer RT, Mbaya OT, Zhou Y, Ploquin A, Sullivan NJ, Graham BS, Roman F, De Ryck I, Ballou WR, Kieny MP, Moorthy V, Spertini F, Genton B. Safety and immunogenicity of a chimpanzee adenovirus-vectored Ebola vaccine in healthy adults: a randomised, double-blind, placebo-controlled, dose-finding, phase 1/2a study. Lancet Infect Dis. 2016 Mar;16(3):311-20. doi: 10.1016/S1473-3099(15)00486-7. Epub 2015 Dec 23. PMID 26725450